CLINICAL TRIAL: NCT00508066
Title: Continuous Local Infusion of Anesthetic at the Incisional Site for Scoliosis Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shriners Hospitals for Children (Other)
Responsible Party: Principal Investigator, Terri Green, Clinical Data Coordinator, Shriners Hospitals for Children
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SHCLA-0116
Record Dates: First submitted 2007-07-25; First posted 2007-07-27 (Estimated); Last update posted 2013-01-25 (Estimated); Status verified 2013-01

CONDITIONS: Scoliosis
Keywords: Congenital Scoliosis; Idiopathic Scoliosis; Spinal Fusion; Post-Operative Pain Management; Infusion Catheter
MeSH Terms: conditions — Scoliosis | interventions — Bupivacaine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental): Subjects in arm 1 will intraoperatively have a continuous infusion catheter placed in the paraspinal musculature of the posterior spinal wound. Post-operatively, the catheter will infuse 0.25 - 0.5% (according to patient's weight) Bupivacaine at a rate of 4ml/hr for 72 hours. This is in addition to the standardized PCA pain management.
  Interventions: Drug: Bupivacaine
- Arm 2 (Placebo Comparator): Subjects in arm 2 will intraoperatively have a continuous infusion catheter placed in the paraspinal musculature of the posterior spinal wound. Post-operatively, the catheter will infuse normal saline at a rate of 4ml/hr for 72 hours. This is in addition to the standardized PCA pain management.
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Drug: Bupivacaine — Bupivacaine 0.25 - 0.5% @ 4ml/hr for 72 hours
  Other Names: Marcaine
  Arms: Arm 1
Drug: Normal Saline — Normal Saline, 4ml/hour for 72 hours.
  Arms: Arm 2

SUMMARY:
The purpose of this study is to evaluate the effects of continuous local anesthetic delivery on the immediate post-op recovery of patients undergoing spinal fusion surgery for congenital or idiopathic scoliosis.

DETAILED DESCRIPTION:
Constant local analgesic infusion is a relatively new modality that provides a constant supply of medication without the need for repeat injections. This method has shown encouraging results with respect to pain levels, narcotic use, faster rehabilitation and shorter hospital stay in patients undergoing laparotomies, iliac crest bone graft harvest, and sternotomies. In addition, there have not been any reported complications when used in these scenarios.

We hope to confirm better pain control, less narcotic use (i.e. PCA), fewer narcotic side effects, better response to physical therapy and earlier discharge. Which may be generalized to the spinal surgery patient population as less pain and suffering and a better overall hospital course

ELIGIBILITY:
Inclusion Criteria:

* Clinical Diagnosis of Congenital Scoliosis
* Clinical Diagnosis of Idiopathic Scoliosis
* Anticipated Spinal Fusion Surgery

Exclusion Criteria:

* Less than 8 years of age

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2007-05; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
VAS pain score | 72 hours

SECONDARY OUTCOMES:
Physical Therapy Progress | Post-op day 1, 2, 3

CONTACTS AND LOCATIONS:
Overall Officials: Norman Otsuka, MD, Study Director — Shriners Hospitals for Children - Los Angeles; Anthony Scaduto, MD, Principal Investigator — Shriners Hospitals for Children - Los Angeles
Locations (1):
- Shriners Hospitals for Children - Los Angeles, Los Angeles, California, United States